CLINICAL TRIAL: NCT07357441
Title: A Retrospective Chart Review Study to Evaluate the Demographics and Treatment Patterns of Myelofibrosis in Routine Practice After Ruxolitinib Approval in Turkey
Brief Title: A Study to Evaluate the Demographics and Treatment Patterns of Myelofibrosis Patients Treated With Ruxolitinib in Turkey
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CINC424ATR01
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Myelofibrosis
Keywords: Real life; Retrospective; Chart review
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Ruxolitinib Group 1: Patients diagnosed with intermediate-1 risk MF according to the Dynamic International Prognostic Scoring System Plus (DIPSS+) at the initial visit who were treated with ruxolitinib.
- Ruxolitinib Group 2: Patients diagnosed with intermediate-2 and High risk MF according to the DIPSS+ at the initial visit who were treated with ruxolitinib.

SUMMARY:
This was a non-interventional retrospective study. Data from patients who were diagnosed with myelofibrosis (MF) (primary MF, post-polycythemia vera MF & post-essential thrombocythemia MF) and treated with ruxolitinib for at least 3 months collectively were collected. The baseline visit was the visit that the patient started ruxolitinib treatment. Data was collected between January 01, 2015 and December 31, 2022. The main baseline clinical and laboratory data of the cohort with at least 3 months of ruxolitinib treatment was documented in order to identify real life patient data in Turkey.

All the data was transferred to a clinical report form (CRF), then to the Statistical Package for the Social Sciences (SPSS) software in an anonymous fashion. The source documents were secured for quality control of the data. The quality control of the data was controlled by an unbiased data entry coordinator.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MF
* Treated with ruxolitinib for at least 3 months

Exclusion Criteria:

None identified.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This was a retrospective, non-interventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Age | Baseline
Number of Patients by Gender | Baseline
Number of Patients by Clinical Characteristic Category | Baseline
  Clinical characteristics included:
  * Janus Kinase (JAK) mutation (yes/no)
  * MF-relevant type of mutation
  * MF Type
  * Cytogenic risk assessment (favorable/unfavorable karyotype)
Time From Diagnosis to Initiation of Ruxolitinib | Baseline
Number of Patients by DIPSS+ Risk Stratification | Baseline, Month 12
  DIPSS+ is a prognostic scoring system used to assign MF patients into 1 of 4 risk categories based on the 8 risk factors: age, hemoglobin level, leukocyte count, percentage of circulating blast cells, presence of constitutional symptoms, platelet count, need for red blood cell transfusion, and unfavorable karyotype. The 4 risk categories are as follows:
  * Low risk (0 points)
  * Intermediate-1 risk (1 point)
  * Intermediate-2 risk (2-3 points)
  * High risk (4-6 points)
Percentage of Patients With Blood Transfusions | Baseline, Month 3, 6, and 12
Percentage of Patients With Splenomegaly | Baseline, Month 3, 6, and 12
Change From Baseline in Percentage of Patients With Splenomegaly | Baseline, Month 12
Percentage of Patients Categorized by Spleen Size | Baseline, Month 3, 6, and 12
  Spleen size was categorized as follows:
  * 20 centimeters (cm) or smaller
  * Bigger than 20 cm
Hemoglobin Levels | Baseline, Month 3, 6, and 12
Hematocrit Levels | Baseline, Month 3, 6, and 12
White Blood Cell (Leukocyte) Count | Baseline, Month 3, 6, and 12
Platelet Count | Baseline, Month 3, 6, and 12
Lactate Dehydrogenase (LDH) Levels | Baseline, Month 3, 6, and 12

SECONDARY OUTCOMES:
Number of Patients With Hematological and Non-hematological Adverse Events | Up to 12 months
Percentage of Patients With Anemia and Thrombocytopenia | Baseline, Month 3, 6, and 12
Percentage of Patients With Treatment Adjustments due to Anemia and Thrombocytopenia | Month 3, 6, and 12
  Treatment adjustments included dose modification, treatment interruption, and treatment discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States